CLINICAL TRIAL: NCT00476606
Title: Treatment Outcome of Children With HIV Infection
Brief Title: A Prospective Cohort of Children With HIV Infection
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Khon Kaen University (Other)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 015
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: HIV children; HAART; ARV; Second line HAART; Viral Load; Combination drug; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Stavudine; Didanosine; Lamivudine; Nevirapine; efavirenz; Saquinavir; Indinavir; Ritonavir; Nelfinavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Long-term pediatric cohort: Long-term follow-up cohort since 2003
  Interventions: Drug: Zidovudine, Stavudine, Didanosine, Lamivudine; Drug: Nevirapine, Efavirenz; Drug: LPV/r, Saquinavir, Indinavir, Ritonavir, Nelfinavir

INTERVENTIONS:
Drug: Zidovudine, Stavudine, Didanosine, Lamivudine — Refer to the Thai guideline for HIV management 2007
Drug: Nevirapine, Efavirenz — Refer to the Thai guideline for HIV management 2007
Drug: LPV/r, Saquinavir, Indinavir, Ritonavir, Nelfinavir — Refer to the Thai guideline for HIV management 2007

SUMMARY:
To evaluate clinical and immunological outcome of children treated with HAART.

DETAILED DESCRIPTION:
This is a long term cohort study that was started in 2002. Currently, there are 120 children enrolled in the study and are receiving HIV care according to standard practice set by the Thai Ministry of Public Health. HIV-infected parents also receive care at the same clinic.

ELIGIBILITY:
Inclusion Criteria:

* Children who are part of the ATC program at Chulalongkorn hospital and at HIV-NAT, The Thai Red Cross AIDS research center
* Children who fulfil criteria to start HAART according to the ATC program
* Children who are switched to second regimen or salvage therapy
* Children who are on any antiretroviral regimens, including post trial children from other HIV-NAT study (both at HIV-NAT and Khon Kaen University sites)
* Children with HIV infection who are not on antiretroviral therapy
* Caretakers understand the purpose of data and plasma samples collection, and have signed the consent form

Exclusion Criteria:

* Patients and caretakers may choose to stop HAART at anytime during the study. If they agree, we would continue to follow them in this study.

Ages: 1 Day to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-infected infants, children and adolescents (range age 1 day - 20 years old) who have participated in HIV-NAT trials
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
1. To collect clinical and immunologic data of children treated with HAART 2. To collect clinical outcome data on children with HIV infection 3. To provide the best possible care to children with HIV infection | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, MSc, Principal Investigator — HIV-NAT, The Thai Red Cross AIDS Research Centre
Locations (3):
- Thailand (3):
  - HIV-NAT, Bangkok
  - Pediatric infectious diseases section, Chulalongkorn University, Bangkok
  - Khon Kaen University, Khon Kaen

REFERENCES:
- [Result] Bunupuradah T., Puthanakit T., Boonrak P., Butterworth O., Mengthaisong T., Intasan J., Ubolyam S., Kosalaraksa P., Engchanil C., Pancharoen C., Lumbiganond P., Phanuphak P., Ananworanich J., HIV-NAT Pediatric Study Team. Efficacy and safety of non nucleoside reverse transcriptase inhibitor (NNRTI) based highly active antiretroviral therapy (HAART) in Thai children with HIV, poster No. TUPEB128. Poster presented at the 4th International AIDS Society Conference on HIV Pathogenesis, Treatment and Prevention, Sydney, Australia, July 22-25, 2007
- [Result] Bunupuradah T, Puthanakit T, Kosalaraksa P, Kerr S, Boonrak P, Prasitsuebsai W, Lumbiganon P, Mengthaisong T, Phasomsap C, Pancharoen C, Ruxrungtham K, Ananworanich J. Immunologic and virologic failure after first-line NNRTI-based antiretroviral therapy in Thai HIV-infected children. AIDS Res Ther. 2011 Oct 26;8:40. doi: 10.1186/1742-6405-8-40. PMID 22026962
- [Result] Sirikum C, Sophonphan J, Chuanjaroen T, Lakonphon S, Srimuan A, Chusut P, Do TC, Prasitsuebsai W, Puthanakit T, Ananworanich J, Bunupuradah T; HIV-NAT 015 study team. HIV disclosure and its effect on treatment outcomes in perinatal HIV-infected Thai children. AIDS Care. 2014;26(9):1144-9. doi: 10.1080/09540121.2014.894614. Epub 2014 Mar 13. PMID 24625136
- See also: Click here for more information about HIV-NAT 015 — http://www.hivnat.org